CLINICAL TRIAL: NCT03910673
Title: A Phase 1 Safety and Intrapulmonary Pharmacokinetics Study of ZTI-01 (Intravenous Fosfomycin Disodium) in Healthy Adult Subjects
Brief Title: Intravenous Fosfomycin Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0058; HHSN272201300017I
Record Dates: First submitted 2019-03-28; First posted 2019-04-10 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2020-03-13

CONDITIONS: Bacterial Infection; Multiple-drug Resistance; Pathogen Resistance
Keywords: Adults; Fosfomycin Disodium; Healthy; Intrapulmonary; Intravenous; Pharmacokinetics; Phase 1; ZTI-01
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- 2-Hour Group (Experimental): ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 2 hours after start of third infusion dose. n = 6
  Interventions: Drug: Fosfomycin disodium
- 30-Minute Group (Experimental): ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 30 minutes after start of third infusion dose. n = 6
  Interventions: Drug: Fosfomycin disodium
- 5-Hour Group (Experimental): ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 5 hours after start of third infusion dose. n = 6
  Interventions: Drug: Fosfomycin disodium
- 75-Minute Group (Experimental): ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 75 minutes after start of third infusion dose. n = 6
  Interventions: Drug: Fosfomycin disodium
- 8-Hour Group (Experimental): ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 8 hours after start of third infusion dose. n = 6
  Interventions: Drug: Fosfomycin disodium

INTERVENTIONS:
Drug: Fosfomycin disodium — Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.

SUMMARY:
This is a Phase 1, open-label, multiple-dose trial conducted at a single center. The treatment period will consist of three 6 g doses (18 g) of ZTI-01 as a 1-hour intravenous (IV) infusion (+10 minute window). A total of 30 enrolled subjects will be randomized to undergo a single standardized bronchoscopy with bronchoalveolar lavage (BAL) at one of five sampling times. A total of 6 subjects will be assigned to each BAL-sampling time. Up to ten additional enrolled subjects will act as alternates to obtain 30 evaluable subjects. An evaluable subject is defined as a subject who receives all doses of ZTI-01, undergoes BAL at the randomized sampling timepoint with BAL return volume adequate for testing, and undergoes at least the one blood sampling timepoint that is concurrent with the assigned BAL sampling timepoint, with blood sampling volume that is adequate for testing. The objectives of the study are to assess safety and pharmacokinetics (PK) for a multiple dose regimen of IV-infused ZTI-01.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multiple-dose trial conducted at a single center. The treatment period will consist of three 6 g doses (18 g) of ZTI-01 as a 1-hour intravenous (IV) infusion (+10 minute window). A total of 30 enrolled subjects will be randomized to undergo a single standardized bronchoscopy with bronchoalveolar lavage (BAL) at one of five sampling times. A total of 6 subjects will be assigned to each BAL-sampling time. Up to ten additional enrolled subjects will act as alternates to obtain 30 evaluable subjects. An evaluable subject is defined as a subject who receives all doses of ZTI-01, undergoes BAL at the randomized sampling timepoint with BAL return volume adequate for testing, and undergoes at least the one blood sampling timepoint that is concurrent with the assigned BAL sampling timepoint, with blood sampling volume that is adequate for testing. The objectives of the study are to assess safety and pharmacokinetics (PK) for a multiple dose regimen of IV-infused ZTI-01.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy* men and women aged 18-45 years with no clinically significant findings** at Screening and Baseline (Day -1 to Day 1)

   *Healthy is defined by the absence of any medical condition described in the exclusion criteria in a subject with a normal physical exam including vital signs. If the subject has another current, ongoing medical condition, the condition cannot meet any of the following criteria: 1) first diagnosed within 3 months of enrollment; 2) is worsening in terms of clinical outcome in the last 6 months; or 3) involves need for medication.

   **Including findings on medical history, physical exam, vital signs, 12-lead Electrocardiogram (ECG), or clinical laboratory tests.
2. Body Mass Index (BMI) = 18 - 30 kg / m^2, inclusive, and body weight > 50 kg (110 lbs).
3. Females who have been surgically sterilized via bilateral oophorectomy and/or hysterectomy at least 90 days prior to Screening are considered lacking childbearing potential and will be eligible*.

   *Postmenopausal females are not eligible, as the definition of menopause would require age > 45, and all subjects in this study are age < / = 45.
4. Females of childbearing potential must have a negative serum pregnancy test at Screening, a negative urine pregnancy test at Baseline (Day -1 to Day 1), and must use acceptable contraception*.

   *Acceptable contraception methods are restricted to surgical sterilization (bilateral tubal ligation) or successful Essure placement (permanent, non-surgical, non-hormonal sterilization with documented radiological confirmation at least 90 days after the procedure), use of long-acting reversible contraceptive devices (progestin-releasing subdermal implants [Nexplanon and Implanon, Merck], copper intrauterine devices [Paragard, Teva], and levonorgestrel-releasing intrauterine devices [Mirena, Bayer; Skyla, Bayer; Liletta, Allergan/Medicines360]), licensed hormonal products such as injectables or oral contraceptives, barrier methods such as condoms or diaphragms with spermicidal agents, and abstinence from sexual intercourse with a male partner. Subjects must have used the above-listed method for a minimum of 30 days prior to the first dose of study drug and be willing to use the method for at least 30 days after the final dose of study drug.
5. Male subjects* whose partners are of childbearing age or pregnant must be willing to use condoms during the study and through the Day 3 follow-up call.

   *including men who have had vasectomies
6. Able to abstain from alcoholic beverages within 48 hours before Baseline (Day -1 to Day 1) and throughout the Treatment Phase.
7. Able to abstain from caffeine use within 7 days before Baseline (Day -1 to Day 1) and throughout the inpatient period.
8. Willing to remain in Duke Early Phase Research Unit (DEPRU) during the Baseline and Treatment Phases.
9. Have a high probability for compliance and completion of the trial.
10. Sign a dated, witnessed, written Informed Consent Form (ICF).
11. Have adequate venous access for infusions and blood draws.

Exclusion Criteria:

1. Any surgical or medical condition that in the opinion of the investigator could interfere with drug absorption, distribution, metabolism, or excretion.
2. Any surgical or medical condition that in the opinion of the investigator may place the subject at increased risk while participating in the trial.
3. History or presence of cardiovascular disease including coronary artery disease and chronic hypertension (systolic pressure > 140 mmHg or diastolic pressure > 90 mmHg).
4. Abnormal Electrocardiogram (ECG) at screening, as determined by the investigator to be clinically significant.
5. History or presence of renal impairment or chronic renal disease.
6. History or presence of liver disease (Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or total bilirubin above the upper limit of normal).
7. History or presence of chronic pulmonary disease, including asthma, requiring use of medication in the year before screening.
8. History of intolerance or hypersensitivity to phosphonic acid derivative antibiotics or any of its constituents (i.e., oral or intravenous fosfomycin).
9. Have cancer or have a history of cancer within the past 5 years, with the exception of non-melanomatous skin cancer, treated, without evidence of recurrence.
10. Any medical condition that prevents a subject from undergoing bronchoscopy with bronchoalveolar lavage (BAL).
11. Serum creatinine above the upper limit of normal, or estimated creatinine clearance (CrCl) < 60 mL / min as determined by Cockcroft-Gault equation*.

    *Cockcroft-Gault equation where age is in years, weight is in kilograms, and serum Cr is in mg/dL units: Males: CrCl (mL / min) = (140 - age) x Weight / (72 x Cr) Females: CrCl (mL / min) = [(140 - age) x Weight / (72 x Cr)] x 0.85
12. History of regular alcohol consumption within 6 months of Baseline (Day -1 to Day 1)*.

    *History of regular alcohol consumption is defined as an average weekly intake of > 14 drinks for males or > 7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine, or 1.5 ounces (45 mL) of 80 proof distilled spirits.
13. History of > / = 10 pack-years smoking, or history of any nicotine use* in the 6 months before Baseline (Day -1 to Day 1)** or positive urinine cotinine screen at Basline (Day -1 to Day 1).

    *Including cigarettes, pipe, cigar, chewing tobacco, nicotine patch.

    **A positive urine cotinine at screening is allowed if negative at baseline.
14. History of illicit drug use within 6 months of Baseline (Day -1 to Day 1)*.

    *Use of cannabinoids within 1 month of Baseline (Day -1 to Day 1) is excluded, but other use of cannabinoids within 6 months is permitted.
15. Use of any prescription drugs, except acceptable contraception methods listed above, within 30 days of Baseline (Day -1 to Day 1).
16. Involvement in other investigational studies of any type (drugs, devices, procedures) within 30 days of Baseline (Day -1 to Day 1).
17. Blood or blood products donation within 30 days of Baseline (Day -1 to Day 1).
18. Planning egg or sperm donation any time before Day 3 follow-up call.
19. Use of any non-prescription medications, vitamins, consumption > 2 times/week of products containing genuine licorice, caffeine, or dietary or herbal supplements within 7 days of Baseline (Day -1 to Day 1)*.

    *Excluded from this list is intermittent use of acetaminophen at doses < / = 2 g / day. Herbal supplements must be discontinued 7 days before the initial dose of study drug on Day 1.
20. Presence of any acute illness, including febrile illness with temperature > 37.8 degrees Celsius (> 100.0 degrees Fahrenheit), within 7 days of Baseline (Day -1 to Day 1).
21. Currently pregnant or breastfeeding as determined by subject report.
22. Positive tests for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
23. Positive urine drug or positive breathalyzer test for alcohol at Screening or Baseline (Day -1 to Day 1) or positive cotinine at Baseline (Day -1 to Day 1).
24. Weight loss or gain of > 10% within 30 days of Baseline (Day -1 to Day 1).
25. Any laboratory value at screening or enrollment that is Grade 2 or more. A laboratory value that is Grade 1 will be allowed if not considered to be clinically significant by the investigator*.

    *Excluded from this list of permissible Grade 1 laboratory values are (ALT), (AST), or Total bilirubin per Exclusion Criteria 6 and serum creatinine per Exclusion Criteria #11; and serum electrolytes including sodium, potassium, calcium, phosphorus and magnesium.
26. History of infection with SARS-CoV-2 (COVID-19) within 3 months of Baseline (Day -1 to Day 1) or unresolved symptoms of COVID-19.
27. Positive test for SARS-CoV-2 (COVID-19) at Screening or Baseline (Day -1 to Day 1) within 72 hours of admission

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina, United States

REFERENCES:
- [Derived] Boole L, Yang Z, Bergin SP, Tighe RM, Randolph E, Hauser B, Gu K, Ghazaryan V, Wall A, Weigand K, Walter EB, Que LG. Evaluation of the safety profile and intrapulmonary pharmacokinetics of intravenous fosfomycin in healthy adults. Antimicrob Agents Chemother. 2025 Feb 13;69(2):e0139524. doi: 10.1128/aac.01395-24. Epub 2025 Jan 8. PMID 39772650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included healthy male and female adults, aged 18-45 years, inclusive, with body mass index (BMI) 18-30 kg/m2, inclusive, and body weight >50 kg (110 lbs) who met all eligibility criteria. Participants were enrolled between 27JUN2019 and 08DEC2020, and were recruited from the community at large.
Groups:
- 30 Minute BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 30 minutes after start of third infusion dose.
  Fosfomycin disodium: Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.
- 75 Minute BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 75 minutes after start of third infusion dose.
  Fosfomycin disodium: Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.
- 2 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 2 hours after start of third infusion dose.
  Fosfomycin disodium: Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.
- 5 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 5 hours after start of third infusion dose.
  Fosfomycin disodium: Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.
- 8 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium. Bronchoscopy and bronchoalveolar lavage (BAL) performed 8 hours after start of third infusion dose.
  Fosfomycin disodium: Fosfomycin (a phosphonic acid derivative) formulated as a disodium salt.
Period: Overall Study
Arm/Group | 30 Minute BAL | 75 Minute BAL | 2 Hour BAL | 5 Hour BAL | 8 Hour BAL
Started | 7 | 6 | 7 | 13 | 6
Enrolled and Randomized | 6 | 6 | 6 | 6 | 6
Enrolled as Replacement | 1 | 0 | 1 | 7 | 0
Began Infusion of Dose 1 | 7 | 6 | 7 | 13 | 6
Completed Dose 1 | 7 | 6 | 7 | 13 | 6
Completed Dose 2 | 7 | 6 | 7 | 13 | 6
Completed Dose 3 | 6 | 6 | 7 | 12 | 6
Completed All Scheduled Treatment | 6 | 6 | 7 | 12 | 6
Completed All PK Blood Draws | 6 | 6 | 6 | 6 | 6
Completed Bronchoscopy With BAL | 6 | 6 | 6 | 6 | 6
Completed All Plasma Urea Samples | 6 | 6 | 6 | 6 | 6
At Least One PK Blood Draw Concurrent With BAL Timepoint | 6 | 6 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 11 | 6
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population includes all participants who received any amount of ZTI-01 (started the first infusion).
Groups:
- 30 Minute BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
  BAL performed 30 minutes after start of third infusion dose.
- 75 Minute BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
  BAL performed 75 minutes after start of third infusion dose.
- 2 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
  BAL performed 2 hours after start of third infusion dose.
- 5 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
  BAL performed 5 hours after start of third infusion dose.
- 8 Hour BAL: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
  BAL performed 8 hours after start of third infusion dose.
- Total: Total of all reporting groups
Arm/Group | 30 Minute BAL | 75 Minute BAL | 2 Hour BAL | 5 Hour BAL | 8 Hour BAL | Total
Number analyzed (Participants) | 7 | 6 | 7 | 13 | 6 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (6.5) | 31.2 (4.6) | 31.4 (6.8) | 32.3 (6.6) | 30.3 (9.4) | 31.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 7 | 3 | 18
  Male | 4 | 5 | 3 | 6 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 6 | 6 | 6 | 10 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 5 | 2 | 15
  White | 3 | 2 | 2 | 5 | 4 | 16
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 170.26 (10.52) | 173 (8.67) | 163.07 (4.54) | 168.22 (8.44) | 173.28 (8.17) | 169.2 (8.62)
Weight [Mean (Standard Deviation); unit: kg] | 70.64 (11.87) | 73.98 (11.26) | 67.6 (6.14) | 74.96 (12.68) | 75.78 (7.49) | 72.84 (10.59)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.31 (3.35) | 24.6 (2.11) | 25.47 (2.68) | 26.89 (2.99) | 25.27 (2.4) | 25.54 (2.84)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve (AUC 0-8 and AUC 0-inf ) of ZTI-01
Description: Mean and standard deviation (SD) of the AUC 0-8 (h*ug/mL) and AUC 0-inf (h*ug/mL). PK parameters were estimated from the ZTI-01 plasma concentration-time data after Dose 1 (Day 1) and Dose 3 (Day 2) using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for the plasma samples collected during the study. AUC 0-8 was estimated for the plasma concentration data after Dose 1 and Dose 3. AUC 0-inf was estimated for the plasma concentration data after Dose 3 with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 1.5 half-lives, and includes at least 3 timepoints after time to maximum concentration (tmax).
Time Frame: Day 1 to Day 2
Population: The PK population includes the population of evaluable participants. An evaluable participant is defined as a participant who received all doses of ZTI-01, underwent BAL at the randomized sampling timepoint with BAL return volume adequate for testing, and obtained at least one blood sample that was concurrent with the BAL sampling timepoint, with blood sampling volume that was adequate for testing.
  All arms are reported jointly as all received the same dose, following the same dosing schedule.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Groups:
- ZTI-01 All Participants: ZTI-01 administered as 1-hour IV infusions (+10 minute window) given every 8 hours for three doses. Each dose comprised of 200 mL (6 g) of fosfomycin disodium.
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
h*ug/mL
  AUC 0-8, after Dose 1 | 780.9 (112.2)
  AUC 0-8, after Dose 3 | 959.4 (147.5)
  AUC 0-inf, after Dose 3 | 1086.0 (183.3)

2. Primary Outcome: Clearance (CL) of ZTI-01
Description: Mean and SD of the clearance (CL) of ZTI-01 (L/h). The clearance PK parameter was estimated from the ZTI-01 plasma concentration-time data after Dose 3 using Phoenix WinNonlin Non-compartmental analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 1.5 half-lives, and includes at least 3 timepoints after time to maximum concentration (tmax). Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for plasma samples collected during the study. If the amount extrapolated portion of AUC 0-inf was >20%, the estimated CL value was excluded from statistical summaries of the parameter estimates.
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
L/h | 5.69 (1.04)

3. Primary Outcome: Intrapulmonary Pharmacokinetics of ZTI-01
Description: Intrapulmonary pharmacokinetics of ZTI-01 was defined as the percent penetration of lung epithelial lining fluid (ELF) and alveolar macrophages (AMs). The estimate of the percent lung penetration was calculated by dividing the AUC 0-8 of ELF and AM by the AUC 0-8 of plasma fosfomycin. The AUC 0-8 of ELF and AM was calculated using the median result at each BAL sampling timepoint, resulting in a single AUC 0-8 of ELF and AM across all subjects. The AUC 0-8 of plasma fosfomycin was calculated using the median result of the plasma fosfomycin concentrations at the corresponding BAL timepoint.
Time Frame: Day 2
Population: as for outcome 1
Measure: Number; unit: Plasma percent penetration
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
Plasma percent penetration
  ELF: number analyzed (Participants) | 29
  ELF | 31.8
  AM | 17.5

4. Primary Outcome: Maximum Measured Plasma Concentration (Cmax) of ZTI-01
Description: Mean and standard deviation (SD) of the Cmax (ug/mL) PK parameter were estimated from the ZTI-01 plasma concentration-time data after Dose 1 and Dose 3 using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for the plasma samples collected during the study.
Time Frame: Day 1 to Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
ug/mL
  Cmax, after Dose 1 | 297.5 (46.074)
  Cmax, after Dose 3 | 335.1 (63.5872)

5. Primary Outcome: Number of Participants Experiencing Abnormal Clinical Chemistry Laboratory Assessments
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Clinical chemistry assessments with toxicity grading and associated thresholds include sodium <135 mEq/L or >145 mEq/L, potassium <3.5 mEq/L or >5.0 mEq/L, random glucose <=69 mg/dL or >=141 mg/dL, blood urea nitrogen (BUN) >=21 mg/dL, creatinine >1.0 mg/dL (Females) or >1.3 mg/dL (Males), calcium <8.7 mg/dL or >10.2 mg/dL, magnesium <=1.7 mg/dL, phosphorous <=2.2 mg/dL, creatine phosphokinase (CPK) >=221 mg/dL, albumin >=2.8 g/dL, total protein <5.8 g/dL, alkaline phosphatase (ALP) >=111 U/L, aspartate aminotransferase (AST) >=42 U/L, alanine aminotransferase (ALT) >54 U/L (Females) or >63 (Males) U/L, total bilirubin >=1.6 mg/dL, direct bilirubin >=0.7 mg/dL, total cholesterol >=301 mg/dL, triglycerides >500 mg/dL, and lactate dehydrogenase (LDH) >200 U/L.
Time Frame: Day 1 to Day 2
Population: The safety population includes all participants who received any amount of ZTI-01 (started the first infusion).
  All arms are reported jointly as all received the same dose, following the same dosing schedule
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Sodium - Increase | 2
  Sodium - Decrease | 2
  Potassium - Increase | 19
  Potassium - Decrease | 19
  Magnesium - Decrease | 31
  Calcium - Increase | 16
  Calcium - Decrease | 16
  Phosphorus - Decrease | 5
  Albumin - Decrease | 4
  Random Glucose - Increase | 8
  Random Glucose - Decrease | 8
  Blood Urea Nitrogen - Increase | 4
  Total Protein - Decrease | 2
  Creatinine - Increase | 0
  Triglycerides - Increase | 5
  Total Cholesterol - Increase | 0
  Creatine Phosphokinase - Increase | 3
  Alkaline Phosphatase - Increase | 1
  Aspartate Aminotransferase - Increase | 0
  Alanine Aminotransferase - Increase | 14
  Total Bilirubin - Increase | 1
  Direct Bilirubin - Increase | 5
  Lactate Dehydrogenase - Increase | 0

6. Primary Outcome: Number of Participants Experiencing Abnormal Clinical Hematology Laboratory Assessments
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Clinical hematology assessments with toxicity grading and associated threshold include hemoglobin <=11.9 g/dL (Females) or <= 13.6 g/dL (Males), white blood cell count <=3.1 10^9/L or >=9.9 10^9/L, lymphocytes <0.6 10^9/L, neutrophils <2.0 10^9/L, eosinophils >0.7 10^9/L, and platelets <=149 10^9/L.
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Hemoglobin - Decrease | 7
  Platelets - Decrease | 1
  WBC - Increase | 7
  WBC - Decrease | 7
  Neutrophils - Decrease | 6
  Lymphocytes - Decrease | 0
  Eosinophils - Increase | 1

7. Primary Outcome: Number of Participants Experiencing Abnormal Clinical Coagulation Laboratory Assessments
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Clinical coagulation assessments with toxicity grading and associated threshold include prothrombin time (PT) >13.1 seconds and activated partial thromboplastic time (aPTT) >37.1 seconds.
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  PT - Increase | 9
  aPTT - Increase | 6

8. Primary Outcome: Number of Participants Experiencing Abnormal Clinical Urinalysis Laboratory Assessments
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Clinical urinalysis assessments with toxicity grading and associated threshold include protein >= 1+, glucose >= 1+, and red blood cell (RBC) count from microscopy >= 5 rbc/hpf.
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Protein | 2
  Glucose | 1
  RBC Count | 1

9. Primary Outcome: Number of Participants Experiencing Abnormal Physical Examination Findings
Description: Physical exams included assessment of skin, head and neck, lungs, heart, liver, spleen, extremities, lymph nodes, musculoskeletal system/extremities, abdomen, nervous system, weight, height, and body mass index (BMI).
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Abdomen | 2
  Extremities | 3
  General Appearance | 4
  Musculoskeletal | 1
  Skin | 2

10. Primary Outcome: Number of Participants Experiencing Abnormal Vital Sign Measurements
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. Vital sign measurements with toxicity grading and associated threshold include systolic blood pressure (BP) >=141 mmHg or <=89 mmHg; diastolic BP >=91 mmHg; heart rate >=101 beats per minute (bpm) and >25% change from baseline or <=54 bpm (if baseline >=60 bpm) or <=49 bpm (if baseline <60 bpm); respiratory rate >=23 breaths per minute; and temperature >=38.0 degrees Celsius.
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Systolic Blood Pressure - Decrease | 2
  Systolic Blood Pressure - Increase | 3
  Diastolic Blood Pressure - Increase | 2
  Heart Rate - Decrease | 13
  Heart Rate - Increase | 6
  Respiratory Rate - Increase | 9
  Temperature - Increase | 0

11. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants who experienced at least one unsolicited treatment emergent AE (TEAE) of any severity and relatedness by MedDRA System Organ Class (SOC). AEs included local and systemic reactions. Any medical condition that was present at screening was considered as a baseline finding and not reported as an AE. However, if its Grade increased at any time during the trial such that it met the AE definition, it was recorded as an AE.
Time Frame: Day 1 to Day 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  Cardiac disorders | 15
  Gastrointestinal disorders | 9
  General disorders and administration site conditions | 10
  Investigations | 37
  Musculoskeletal and connective tissue disorders | 1
  Nervous system disorders | 5
  Renal and urinary disorders | 1
  Respiratory, thoracic and mediastinal disorders | 14
  Skin and subcutaneous tissue disorders | 2
  Vascular disorders | 7

12. Primary Outcome: Number of Participants With Prolonged QTc, PR, or QRS Intervals in Electrocardiogram (ECG) Readings
Description: Each subject is only counted once per toxicity grade for the worst severity recorded. ECG assessments with toxicity grading and associated threshold include QTc Interval >=450 msec, PR Interval >=200 msec and >25% change from baseline, and QRS Interval >=120 msec and >25% change from baseline.
Time Frame: Day 1 to Day 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 39
Participants
  QTc Interval | 1
  PR Interval | 0
  QRS Duration | 0

13. Primary Outcome: Terminal Elimination Half-life (t1/2) of ZTI-01
Description: Mean and standard deviation (SD) of the t1/2 (h) PK parameter were estimated from the ZTI-01 plasma concentration-time data after Dose 3 using Phoenix WinNonlin Non-compartmental analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 1.5 half-lives, and includes at least 3 timepoints after time to maximum concentration (tmax). Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for the plasma samples collected during the study.
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
h | 2.62 (0.36)

14. Primary Outcome: Terminal-phase Elimination Rate Constant (Lambdaz) of ZTI-01
Description: Mean and standard deviation (SD) of the lambdaz (/h) PK parameter were estimated from the ZTI-01 plasma concentration-time data after Dose 3 using Phoenix WinNonlin Non-compartmental analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 1.5 half-lives, and includes at least 3 timepoints after time to maximum concentration (tmax). Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for the plasma samples collected during the study.
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: /h
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
/h | 0.2703 (0.0391)

15. Primary Outcome: Time to Peak Concentration (Tmax) of ZTI-01
Description: Mean and standard deviation (SD) of the Tmax (h) PK parameter were estimated from the ZTI-01 plasma concentration-time data after Dose 1 and Dose 3 using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for the plasma samples collected during the study.
Time Frame: Day 1 to Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
h
  Tmax, after Dose 1 | 1.07 (0.06)
  Tmax, after Dose 3 | 1.06 (0.05)

16. Primary Outcome: Volume of Distribution at Steady State (Vss) of ZTI-01
Description: Mean and standard deviation (SD) of the Vss (L) PK parameter were estimated from the ZTI-01 plasma concentration-time data after Dose 3 using Phoenix WinNonlin Non-compartmental analysis with the following Lambda Z Acceptance Criteria: rsq_adjusted (adjusted r squared) >= 0.90, span >= 1.5 half-lives, and includes at least 3 timepoints after time to maximum concentration (tmax). Plasma concentrations were measured by a validated LC-MS/MS bioanalytical assay for plasma samples collected during the study. If the amount extrapolated portion of AUC 0-inf was >20%, the estimated Vss value was excluded from statistical summaries of the parameter estimates.
Time Frame: Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | ZTI-01 All Participants
Number analyzed (Participants) | 30
L | 18.08 (2.80)

ADVERSE EVENTS:
Time Frame: The period of observation for AE reporting began on Day 1 at the time of first dosing and continued through the final visit, a follow-up call on Day 3.
Arm/Group | ZTI-01 All Participants
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 38/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZTI-01 All Participants (N=39)
Bradycardia (Cardiac disorders) | 7 (8)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Infusion site pain (General disorders) | 3 (3)
Vessel puncture site pain (General disorders) | 2 (2)
Blood albumin decreased (Investigations) | 3 (3)
Blood calcium decreased (Investigations) | 16 (16)
Blood glucose increased (Investigations) | 7 (7)
Blood magnesium decreased (Investigations) | 29 (29)
Blood phosphorus decreased (Investigations) | 4 (4)
Blood potassium decreased (Investigations) | 19 (19)
Haemoglobin decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 3 (3)
Protein urine present (Investigations) | 2 (2)
Prothrombin time prolonged (Investigations) | 6 (6)
White blood cell count decreased (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Diastolic hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Systolic hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03910673/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03910673/SAP_002.pdf
  • Informed Consent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03910673/ICF_000.pdf